CLINICAL TRIAL: NCT01898351
Title: Health Impacts of Sustainable Ingredient Selection in the Food and Drink Industry - ALTERNATIVE PROTEIN STUDY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aberdeen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Alternative Protein Study 791
Record Dates: First submitted 2013-07-09; First posted 2013-07-12 (Estimated); Last update posted 2015-11-13 (Estimated); Status verified 2015-11

CONDITIONS: Healthy
Keywords: Alternative sources of plant proteins; High protein diets; Satiety; Postprandial effects; Bioactive phytochemicals; Phytochemicals bioactivity and metabolism; Macronutrients metabolism; Health effects of plant proteins vs. meat proteins; Partial meat proteins replacement with plant proteins; Satiety of meals rich in plant proteins; Postprandial effects of meals rich in plant proteins; Plant phytochemicals and macronutrients bioavailability and metabolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fava bean, Lupin, Beef meat, Green pea, Hemp, Buckwheat (Other): The intervention visit involves a test meal to be consumed by subjects attending the Human Nutrition Unit in the morning, following an overnight fast. The meal will be consumed within 15 minutes and blood (69 mL) and urine samples will be collected during 24 hours.
  The test meals are designed to contain the same amount of proteins. Alternative protein meals: a number of bread buns for each meal containing individual alternative protein flours (green pea, lupin, hemp, buckwheat, fava beans). These will deliver 30 g of protein, the remainder being provided by white flour. The control (meat) meal: a lean beef steak containing 30 g of protein and a bun containing the same amount of white flour as used for the alternative protein bread buns.
  The semi structured interview guide: will take place within the Human Nutrition Unit during one of the scheduled visits, once initial screening has taken place and participants have been selected. All interviews will be digitally recorded.
  Interventions: Other: Fava bean, Lupin, Beef meat, Green pea, Hemp, Buckwheat

INTERVENTIONS:
Other: Fava bean, Lupin, Beef meat, Green pea, Hemp, Buckwheat — The intervention visit involves a test meal to be consumed by subjects attending the Human Nutrition Unit in the morning, following an overnight fast. The meal will be consumed within 15 minutes and blood (69 mL) and urine samples will be collected during 24 hours.
  The test meals are designed to contain the same amount of proteins. Alternative protein meals: a number of bread buns for each meal containing individual alternative protein flours (green pea, lupin, hemp, buckwheat, fava beans). These will deliver 30 g of protein, the remainder being provided by white flour. The control (meat) meal: a lean beef steak containing 30 g of protein and a bun containing the same amount of white flour as used for the alternative protein bread buns.
  The semi structured interview guide: will take place within the Human Nutrition Unit during one of the scheduled visits, once initial screening has taken place and participants have been selected. All interviews will be digitally recorded.

SUMMARY:
Summary

This research will examine the nutritional effects of supplementing diets with alternative plant sources of protein with potential to be grown in Scotland. In particular, we will assess the potential of these plant protein sources to complement diets in which the predominant source of protein is meat. These protein sources will include plants from the Fabaceae, Cannabaceae and Polygonaceae families, which could be used as the basis for the development of new foods. The research will assess if these plant proteins can deliver a comparable alternative to meat based diets.

It is anticipated that the results could encourage increased consumption of plant products which would be favorable for consumers shifting away from animal-derived proteins for health and/or environmental reasons.

Hypothesis: Consumption of protein rich plants could be a sustainable and healthy choice for partial replacement in predominantly meat based diets.

Objective: The objective of this acute study is to assess satiety, postprandial effects, metabolite bioavailability and metabolism of single alternative proteins from a shortlist including buckwheat, fava beans, lupin, pea, and hemp in comparison with red meat.

Study protocol

Aims: To assess the impact of a pea, fava bean, lupin, hemp, buckwheat in comparison with meat in healthy people on:

* Biomarkers of satiety as measured by gut-related hormones and subjective appetite using visual analogue scales, specifically to be collected during the meal over a three hour period, every 30 minutes. The energy intake measured for each volunteer after an ad libitum lunch (five hours after test meal).
* Biomarkers of CVD risk including total cholesterol, low density lipoproteins (LDL), high density lipoproteins (HDL), triglycerides and non-esterified fatty acids (NEFA).
* Assessment of peripheral glycaemic control, fasting glucose, area under the curve combined with insulin data.
* Plasma and urine markers of important phytochemical and protein metabolites will be quantitatively analysed to determine the systemic availability, in vivo concentrations and excretion times.
* Volunteer views towards diets rich in plant proteins will be assessed.

DETAILED DESCRIPTION:
Background

Recent scientific evidence suggests that diets largely based on plant foods, such as well-balanced vegetarian diets, have potential to improve health, in contrast with predominantly meat-based diets. However, many consumers may not wish to exclude meat from the diet, despite current advice to reduce, in particular, processed meat. One way to achieve this is to increase consumption of plant-based protein components in the diet.

Making a comparison of the nutritional content of high protein plants (i.e. those with > 20 g protein/100 g dry weight), several candidate sources were identified. In particular, these belong to the Fabaceae family and include pulses (green peas, fava beans, lupin seeds) and certain common bean species. Species from plant families other than the Fabaceae generally have less protein. An exception is hemp seed (Cannabaceae family), which can have a protein content around 40g protein /100g dry weight, is a source of fibre, and has favourable fatty acid and amino acid profiles. Other families of interest include the Amaranthaceae species (Quinoa), Polygonaceae (Buckwheat) and the Poaceae (Wheat, Barley and Oats). Protein content of these pseudocereal and cereal crops ranges from 12-20 g protein /100 g dry weight. Although lower in protein content compared with the Fabaceae species, they are generally rich in fibre and consequently will impart additional benefits to a high-protein plant based diet.

According to the Scottish Health Survey (2009), nearly two-thirds of men (66.3%) and approximately half of women (58.4%) were overweight. Obesity is a major risk factor for metabolic syndrome, which is linked to conditions such as type II diabetes mellitus (T2DM). Having impaired glucose tolerance doubles the chance of morbidity and mortality from cardiovascular disease (CVD). CVD is the leading cause of death and accounts for nearly 30% of deaths worldwide each year. Clinical studies have shown that regular consumption of pulses can reduce blood levels of total cholesterol and low density lipoprotein (LDL).

The recent meta-analysis of randomized controlled trials provides the strongest evidence to date that non-soya legume consumption lowers serum total and LDL cholesterol and therefore, may lower the risk of CVD. Eating pulses regularly may also lower CVD risk via favorable effects on blood pressure, blood glucose and insulin levels and by satisfying hunger and helping manage body weight. Higher legume intakes were associated with lower body mass index (BMI), blood pressure, serum total cholesterol (TC) and a lower incidence of T2DM, compared with lower legume intakes. In addition to achieving energy balance and improving the overall diet, the World Health Organization (WHO) recommends that people increase consumption of legumes (pulses), as well as vegetables, wholegrain and nuts to prevent obesity. There does not seem to be differential effects of pea-protein as compared to other meat and dairy proteins when fed at similar amounts as a pre-load.

Technically a nut, hempseed typically contains over 30% oil and about 25% protein, with considerable amounts of dietary fibre, vitamins and minerals. The two main proteins in hempseed are edestin and albumin (high-quality storage proteins are easily digested and contain nutritionally significant amounts of all essential amino acids); hempseed has exceptionally high levels of the amino acid arginine. Hempseed is an excellent source of nutrition and has been used to treat various disorders for thousands of years in traditional medicine. Animal studies and only few humans study (on hemp seeds oil) agree as well that hempseed has health promoting properties; supported by results from nutritional analyses of the seed, oil and seed meal. Being a rich source of polyunsaturated fatty acids and proteins which contain all of the essential amino acids in nutritionally sufficient amounts as detailed by the FAO/WHO (Food and Agriculture Organization of the United Nations/World Health Organization) suggested requirements for infants or children. Hemp proteins have a Protein Digestibility Corrected Amino Acid Score (PDCAAS) equal to or greater than certain grains, other nuts, and some pulses. Hempseed, in addition to its nutritional value, has demonstrated positive health benefits, including the lowering of cholesterol and high blood pressure.

Buckwheat has attracted increasing attention from food scientists for its potential beneficial effects in chronic diseases. In the early 1970's the nutritional properties of buckwheat were first demonstrated. The cholesterol lowering effects of buckwheat protein extracts in rats with cholesterol-enriched diets has been reported.

There has been much research conducted on the functionalities and properties of buckwheat proteins and other phytochemicals in buckwheat seeds. Among them, the most promising are the flavones, flavonoids, phytosterols, fagopyrins, and the thiamin-binding proteins. Buckwheat proteins have unique amino acid compositions Experiments, both in animal models and with human studies revealed that buckwheat flour can improve T2DM, obesity, hypertension, hypercholesterolemia and constipation.

For the social science element of the project, the proposed study will employ qualitative research methods which emphasise the importance of 'lay' knowledge and the subjective experience of research participants. Within the field of nutrition research, qualitative methods and techniques still remain comparatively rare. This is partly because of the privileged status of quantitative research, but also because of the length of time and amount of effort that goes into each qualitative study and the small pool of qualified researchers in this field .As qualitative research efforts require that researchers seek to understand people and the social and cultural contexts in which they live from the participants' points of view, this type of knowledge has much to contribute to our understanding of why people eat what they do. For the purposes of this study, qualitative methods will enhance our understanding of the acceptability, to consumers in Scotland, of foods based on sustainable, plant-based protein. It will also tell us much about any barrier that exist to the uptake of such foods, from a consumer perspective.

Planned work for the study

From a health perspective it is essential to establish the bioavailability and metabolism of plant proteins and other dietary constituents in humans. Certain metabolites are absorbed early in the gastrointestinal tract, whereas others are transported to the colon where they are extensively metabolized by the gut microbiota. In this acute study, we will characterise the bioactive metabolites present in the urine and plasma samples obtained. This will inform on their availability to the systemic circulation, as well as their excretion profiles. We will employ targeted quantitative analysis using both LC-MS and GC-MS which will provide the identity of metabolites and their in vivo concentrations. We will focus on metabolites that are considered to impact on human health. The principal metabolites analysed will be those produced by the phenylpropanoid pathway and products of protein and carbohydrate metabolism. These will include derivatives and metabolites of the simple phenols, benzoic acids, phenolic acids, phenylacetic acids, phenypropionic acids, phenylpyruvic acids, phenyllactic acids, mandellic acids, phenolic dimers, acetophenones, benzaldehydes, cinnamaldehydes, benzyl alcohols, cinnamyl alcohols, indoles, isoflavones, coumarins, chalcones, flavanones, flavones, flavonols, anthocyanidins. We have also shown that many of these compounds are bioactive and exhibit anti-oxidant and anti-inflammatory activity at in vivo concentrations. These studies will provide important information on bioavailability and metabolism, but will also allow us to correlate the indices with biomarkers of health. In this study we will also examine the effect of different protein sources on post-prandial effects, endocrine responses (e.g. PYY (peptide YY) levels) and hunger ratings. The energy intake for each volunteer will be measured after lunch (ad libitum) on the intervention day. Volunteer views and acceptability towards diets rich in plant protein will be assessed. Some components in pulses may contribute to weight control by inhibiting intestinal absorption of carbohydrates and other energy yielding nutrients such as protein. Correlating the metabolic profiles with biomarkers of health will provide information that will be fed back into agricultural practice to optimise crop breeding strategies for benefits on human health.

With regard to the social science component of the project, in-depth semi-structured interviews will be used. The term 'semi-structured' reflects the intrinsic flexibility of qualitative interview approaches, which often use an aide-memoire or interview guide rather than a formal schedule. In addition, the form and content of the research questions is likely to vary, in response to each particular interview context. This type of built-in design can strengthen qualitative research because of its attentiveness to context.

All interviews will be digitally recorded and fully transcribed. The qualitative analytical techniques applied will look for and examine the themes and patterns of meaning within the kinds of data generated by this research mode. The interviews and conversations that take place as part of qualitative inquiry will generate responses, perceptions, opinions and so on from research participants. These can be understood as constituting a 'discourse' (or set of ideas) derived from the focus of the inquiry that lends itself particularly well to thematic analysis. Themes are derived by the process known as 'coding' (or labelling) specific chunks of text according to the ideas which they seem to represent. This interpretative work involves the creation of analytical themes by the researcher and is particularly useful in bringing together the 'insider' or 'emic' perspective derived from the research participant's knowledge and experience, with the 'outsider' or 'etic' perspective of the researcher and the relevant literature. Patterns in the data are thus identified through the intellectual work of bringing together components or fragments of ideas, perceptions or experiences which might be meaningless when considered in isolation. The researcher engaged in thematic analysis seeks to understand how different ideas or components fit together in a meaningful way, in order to produce a coherent analytical account.

The analysis will be validated by referring back to the relevant literature, which may support (or counter) inferences drawn by the researcher. The interweaving of research findings with extant research literature will help strengthen the interpretive account provided by the researcher. Research participants will also be engaged in this process in that their feedback on emerging patterns will be sought. This process of member checking will be conducted during the course of each interview. Through an analytical framework that focuses on discourse and acknowledges the importance of participants' own perspectives and experiences, analysis will present a contextualised exploration of the ways in which consumers perceive plant-based proteins as alternatives or supplements to meat.

ELIGIBILITY:
Inclusion Criteria:

Healthy males and females, non-vegetarians, non-smokers, age 18-65 with BMI 18-35 kg m-2, taking no exclusion criteria medication.

Exclusion Criteria:

Diabetes Severe gastrointestinal disorders Kidney disease Thromboembolic or coagulation disease Hepatic disease Alcohol or any other substance abuse Gout Eating disorders Allergy Unregulated thyroid disease Asthma Eczema Hay fever Gluten/wheat intolerance Psychiatric disorder resulting in a perceived inability to give informed consent (including severe depression, lithium treatment, schizophrenia, severe behavioral disorders)

Medication exclusion criteria (Confirmed with GP) Orlistat (Xenical) Oral antidiabetics, insulin Digoxin, anti-arrhythmics Anti-inflammatories/anti-pyretics Tricyclic antidepressants, neuroleptics Antihistamines

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-03; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Postprandial effects (including satiety )of a pea, fava bean, lupin, hemp, buckwheat in comparison with meat in healthy people. | up to 3 months
  Each intervention visit will involve a test meal to be consumed by subjects attending the Human Nutrition Unit (HNU) in the morning, following an overnight fast. They will be provided with a meal, which will be consumed within 15 minutes and blood (69 mL) and urine samples will be collected during 24 hours .
  Biomarkers of satiety as measured by gut-related hormones and subjective appetite using visual analogue scales, specifically to be collected during the meal over a three hour period, every 30 minutes. The energy intake measured for each volunteer after an ad libitum lunch (five hours after test meal).
  Biomarkers of CVD risk including total cholesterol, low density lipoproteins (LDL), high density lipoproteins (HDL), triglycerides and non-esterified fatty acids (NEFA).
  Assessment of peripheral glycaemic control, fasting glucose, area under the curve combined with insulin data.

SECONDARY OUTCOMES:
Metabolite bioavailability and metabolism of single alternative proteins from a shortlist including buckwheat, fava beans, lupin, pea, and hemp in comparison with red meat. | up to 3 months
  The intervention visit will involve a test meal to be consumed by subjects attending the Human Nutrition Unit (HNU) in the morning, following an overnight fast. They will be provided with a meal, which will be consumed within 15 minutes and blood (69 mL) and urine samples will be collected during 24 hours
  Plasma and urine markers of important phytochemical and protein metabolites will be quantitatively analysed to determine the systemic availability, in vivo concentrations and excretion times.

OTHER OUTCOMES:
Volunteer views towards diets rich in plant proteins will be assessed. | The assesment will take place during one of the interventtion visits of the study and will be around one hour long.
  With regard to the social science component of the project, in-depth semi-structured interviews will be used for assessing the volunteers view towards diets rich in alternative plant proteins. For each volunteer will be conducted an digitally recorded interview(one hour), during one of the scheduled visits at the Human Nutrition Unit, once initial screening has taken place and participants have been selected.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra M Johnstone, PhD, Principal Investigator — Rowett Institute of Nutrition and Health, University of Aberdeen, Scotland, UK; Madalina Neacsu, PhD, Principal Investigator — Rowett Institute of Nutrition and Health, University of Aberdeen, Scotland, UK; Wendy R Russell, PhD, Principal Investigator — Rowett Institute of Nutrition and Health, University of Aberdeen, Scotland, UK; Sandra Carlisle, PhD, Principal Investigator — Rowett Institute of Nutrition and Health, University of Aberdeen, Scotland, UK
Locations (1):
- Rowett Institute of Nutrition and Health, University of Aberdeen, Aberdeen, Scotland, United Kingdom

REFERENCES:
- [Derived] Neacsu M, Vaughan NJ, Multari S, Haljas E, Scobbie L, Duncan GJ, Cantlay L, Fyfe C, Anderson S, Horgan G, Johnstone AM, Russell WR. Hemp and buckwheat are valuable sources of dietary amino acids, beneficially modulating gastrointestinal hormones and promoting satiety in healthy volunteers. Eur J Nutr. 2022 Mar;61(2):1057-1072. doi: 10.1007/s00394-021-02711-z. Epub 2021 Oct 30. PMID 34716790